CLINICAL TRIAL: NCT03133741
Title: Inhibition of the Endogenous GIP Response With a GIP Receptor Antagonist (GA-3)
Brief Title: Inhibition of the Endogenous GIP Response With a GIP Receptor Antagonist
Acronym: GA-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lærke Smidt Gasbjerg, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UHG-CFD-GIPANTA-3
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Glucose Metabolism Disorders
Keywords: GIP; GIP receptor antagonist
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Sodium Chloride; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo
- GIP-A (Other): Infusion of GIP-A alone as study tool.
  Interventions: Other: GIP-A
- GLP-1 receptor antagonist Exendin[9-39] (Other): Infusion of GLP-1 receptor antagonist Exendin[9-39] alone as study tool.
  Interventions: Other: GLP-1 receptor antagonist Exendin[9-39]
- GIP-A + Exendin[9-39] (Other): Infusion of GIP-A + GLP-1 receptor antagonist Exendin[9-39] together as study tools.
  Interventions: Other: GIP-A + Exendin[9-39]

INTERVENTIONS:
Other: GIP-A — GIP-A (GIP receptor antagonist)
  Arms: GIP-A
Other: GLP-1 receptor antagonist Exendin[9-39] — Exendin[9-39]
  Other Names: EX(9-39)
  Arms: GLP-1 receptor antagonist Exendin[9-39]
Other: Placebo — Saline (9mg/mL)
  Other Names: Saline
  Arms: Placebo
Other: GIP-A + Exendin[9-39] — GIP receptor antagonist + GLP-1 receptor antagonist
  Arms: GIP-A + Exendin[9-39]

SUMMARY:
Delinieation of GIP's effects during an oral glucose tolerance test (OGTT) in humans using GIP receptor antagonisation.

DETAILED DESCRIPTION:
Aim: To evaluate the role of GIPR signalling in postprandial physiology, including bone and glucose homeostasis, using a naturally occurring GIP fragment (GIP-A), which antagonises the GIPR.

Eighteen healthy men (age 18-70 years, BMI 19-35 kg/m2) with normal kidney and liver parameters and haemoglobin levels and no first-degree relatives with type 2 diabetes will be included in a randomised, double-blinded, placebo-controlled cross-over study. Study consists of four study days with concomitant infusions of A) GIP-A, B) GLP-1 receptor antagonist Exendin[9-39], C) GIP-A + Exendin[9-39], or D) saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Normal kidney function, liver function and hemoglobin levels.

Exclusion Criteria:

* Medication, Diabetes type 1 or 2, first degree relatives with Diabetes type 2

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Insulin levels | 240 minutes
  Serum insulin AUC (area under the curve)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — UHGentofte, Center for Diabetes Research
Locations (1):
- Center for Diabetes Research, Gentofte Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Helsted MM, Gasbjerg LS, Lanng AR, Bergmann NC, Stensen S, Hartmann B, Christensen MB, Holst JJ, Vilsboll T, Rosenkilde MM, Knop FK. The role of endogenous GIP and GLP-1 in postprandial bone homeostasis. Bone. 2020 Nov;140:115553. doi: 10.1016/j.bone.2020.115553. Epub 2020 Jul 27. PMID 32730920
- [Derived] Gasbjerg LS, Helsted MM, Hartmann B, Jensen MH, Gabe MBN, Sparre-Ulrich AH, Veedfald S, Stensen S, Lanng AR, Bergmann NC, Christensen MB, Vilsboll T, Holst JJ, Rosenkilde MM, Knop FK. Separate and Combined Glucometabolic Effects of Endogenous Glucose-Dependent Insulinotropic Polypeptide and Glucagon-like Peptide 1 in Healthy Individuals. Diabetes. 2019 May;68(5):906-917. doi: 10.2337/db18-1123. Epub 2019 Jan 9. PMID 30626611